CLINICAL TRIAL: NCT02696213
Title: Systematic, Comprehensive, One-to-One Training (SCOOT) for Scooter Skills: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Mortenson, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H15-01921; F15-00959 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2016-02-23; First posted 2016-03-02 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Mobility Scooter Skills Training

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- SCOOT Immediate (Experimental): This group will receive SCOOT immediately
  Interventions: Other: Systematic, Comprehensive, One to One Training (SCOOT)
- SCOOT Delayed (Other): This group will receive SCOOT after 6 weeks
  Interventions: Other: Systematic, Comprehensive, One to One Training (SCOOT); Other: Six Week Delay

INTERVENTIONS:
Other: Systematic, Comprehensive, One to One Training (SCOOT) — An occupational therapist trained by the principal investigator will perform 1.5 hour SCOOT sessions with participants one to two times a week over a period of 6 weeks. SCOOT will provide instruction and practice for performing scooter skills (i.e., instruction on driving, basic and advanced scooter skills) that are embedded in self-selected activities that participants want to perform using their scooters.
Other: Six Week Delay — Participants will begin the SCOOT intervention after a six week delay.
  Arms: SCOOT Delayed

SUMMARY:
Systematic, Comprehensive, One-to-One Training (SCOOT) for Scooter Skills, is a novel, community-based, client-centred intervention where skills training is incorporated into social activities that users want to perform. The trainer also offers problem solving strategies to help manage environmental barriers and to promote social participation. This intervention is different from customary scooter training in that customary training is often very limited and focuses on learning discrete skills outside of the user's normal environment. The purpose of this study is to explore the feasibility of conducting a mixed-methods, rater-blinded, randomized controlled trial (RCT) for new scooter users, which will evaluate the efficacy of SCOOT. We anticipate that the feasibility outcomes will be strong enough to support the conduct of a subsequent multi-site trial with a sufficient sample size to enable us to quantify definitive outcomes such as adverse events (e.g., injuries and abandonment).

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Aged 60 or above
* Has acquired a scooter in the last month prior to enrollment in the study

Exclusion Criteria:

* Has a cognitive impairment that will prevent the individual from providing consent and reliably completing the study questionnaires
* Reside in a nursing home
* Plan to move outside Vancouver within the next year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Change in scooter skills capacity | Change from baseline skill level at 6 weeks, 12 weeks, 6 months, and 1 year
  The WST-ScQ measures the participant's subjective scooter skills (capacity), and inquires on the frequency the skill is performed, and whether or not improvement of the skill is a personal goal.

SECONDARY OUTCOMES:
Wheelchair Skills Test for Scooters (WST-Sc) | Baseline, at 6 weeks, 12 weeks, 6 months, and 1 year
  The WST-Sc consists of 29 skills that are scored by an examiner from 0 to 2, where 0 = unsafe or unable, 1 = safe with difficulty, and 2 = safe without difficulty
Wheelchair Skills Test for Scooters - Questionnaire (WST-ScQ) (performance and confidence) | Baseline, at 6 weeks, 12 weeks, 6 months, and 1 year
  The WST-ScQ measures the participant's subjective scooter skills, and inquires on the participant's scooter skill confidence, frequency the skill is performed (performance), and whether or not improvement of the skill is a personal goal.
Scooter Skills Confidence Questionnaire | Baseline, at 6 weeks, 12 weeks, 6 months, and 1 year
  This measure evaluates the participant's confidence in managing their social environment
Wheeled Mobility Outcome Questionnaire | Baseline, at 6 weeks, 12 weeks, 6 months, and 1 year
  This measure evaluates indoor and outdoor participation levels associated with wheeled mobility provision by using an 11 point scale (0 = completely unsatisfied to 10 = completely satisfied).
Life Space Assessment (LSA) Questionnaire | Baseline, at 6 weeks, 12 weeks, 6 months, and 1 year
  The LSA measures participants' frequency and independence of mobility in increasingly larger life spaces over the past month.
Scooter Use and Incidents | Baseline, 6 weeks, 12 weeks, 6 months, and 1 Year
  Participants will be asked to keep a diary of any scooter-related adverse events, including the following: tips or falls from the scooter, injuries to self, accidental contact with others, injuries to others, and damage to property. Participants will be asked to record the number of hours per day that they use their scooters.

OTHER OUTCOMES:
Montreal Cognitive Assessment Test | Baseline
  This assessment is used to detect any mild cognitive impairments
Late Life Functioning and Disability measure - Computer Assisted Testing (LLFDI - CAT) | Baseline
  The LLFDI-CAT is a computerized program that measures the participant's physical function. Drawing from a bank of 141 items, CAT continues until a standard error of 3 is obtained for the domain score, or a maximum of ten items has been administered.
Hearing Handicap Inventory for the Elderly (HHIE) Screening version | Baseline
  The HHIE will be used to evaluate the participants' hearing abilities.
Scooter Physical Accessibility of Participant Home and Community | Baseline
  This measure involves 14 yes/no questions inquiring about the accessibility of the participants' physical environment in their home and community.
Trail Making B Test | Baseline
  This task is used to measure the participants' visual attention and task switching abilities, which is related to on road driving
Snellen Eye Test | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ben Mortenson, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Center, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Kirby RL, Smith C, Mortenson WB, Battalova A, Hurd L, Hobson S, Jang S, Emery R. Qualitative experiences of new motorised mobility scooter users relevant to their scooter skills: a secondary analysis. Disabil Rehabil Assist Technol. 2023 Jan;18(1):89-96. doi: 10.1080/17483107.2022.2063422. Epub 2022 Apr 20. PMID 35442822
- [Derived] Mortenson WB, Jang S, Goldsmith CH, Hurd Clarke L, Hobson S, Emery R. Feasibility of a Systematic, Comprehensive, One-to-One Training (SCOOT) program for new scooter users: study protocol for a randomized control trial. Trials. 2017 May 25;18(1):235. doi: 10.1186/s13063-017-1963-y. PMID 28545498